CLINICAL TRIAL: NCT04687930
Title: Genicular Nerve Block in Juvenile Idiopathic Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahrous, Associate professor, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8122020
Record Dates: First submitted 2020-12-19; First posted 2020-12-29 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Juvenile Idiopathic Arthritis; Persistent Knee Arthritis; no Intra-articular Injection in the Last 3 Months; no Other Cause for Chronic Kneearthritis
Keywords: Juvenile rheumatoid arthritis; knee joint; Nerve block
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Steroids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active genicular nerve block group (Active Comparator): group 1 will receive genicular nerve block. The injection and US examination will be done by two experienced sonographers. They were blinded to clinical data. Patients will also be blinded for the injected substance. Each point will be injected with 2 ml of Lidocaine hydrochloride 2 % (Xylocaine, Astrazeneca). The injection will be done using the 3 point technique (superior medial, superior lateral, and inferior medial genicular nerves).
  Interventions: Drug: genicular nerve block
- intra-articular steroid injection group (Other): while group 2 received intra-articular triamcinolone under ultrasound guidance and through injecting the supra-patellar bursa.
  Interventions: Drug: intra-articular steroid injection

INTERVENTIONS:
Drug: genicular nerve block — nerve block of the genicular nerve at 3 points around the inflamed knee using ultrasound.
  Arms: Active genicular nerve block group
Drug: intra-articular steroid injection — Triamcinilone injection into the knee joint under ultrasound guidance.
  Arms: intra-articular steroid injection group

SUMMARY:
N=104 juvenile idiopathic arthritis patients diagnosed after ILAR criteria with unilateral persistent knee arthritis. They will be randomly assigned into two groups; group 1 will receive genicular nerve block, group 2 intra-articular triamcinolone. Both groups will be examined by SOLAR ultrasound scoring system, Visual analogue scale and Lysholm score at 0, 2 and 12 weeks. A semi-quantitative score will be used to assess tenderness and swelling at the same intervals.

ELIGIBILITY:
Inclusion Criteria:

* juvenile idiopathic arthritis with persistent knee arthritis
* age below 16

Exclusion Criteria:

* severe knee osteoarthritis
* peripheral neuropathy,
* psoriatic arthritis,
* those under anticoagulant therapy, skin infection,
* prior knee injection in the last 3 months3
* those who have an allergy to Bupivacaine

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Change in SOLAR score over time | Baseline, 2 weeks and 12 weeks
  score to assess ultrasound parameters of the knee including power doppler and grey scale measures
Change in visual analogue scale over time | Baseline, 2 weeks and 12 weeks
  a graded score for pain evaluation filled by the patient graded from 0 to 10
Change in Lysholm score over time | Baseline, 2 weeks and 12 weeks
  a score to assess knee function. This questionnaire has 8 domains. A score between 95 and 100 means excellent functional performance, good 84-94, fair 65-83 and poor <64
Change in semiquantitative score for swelling and tenderness over time | Baseline, 2 weeks and 12 weeks
  A score graded from 0 to 3; score 0 means no swelling nor tenderness and 3 means maximum swelling and tenderness

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt

REFERENCES:
- [Derived] Radwan A, Ohrndorf S, Aly H, Hamed M, Khalifa A, Elsaman AM. Genicular nerve block in juvenile idiopathic arthritis: a randomized clinical trial. Clin Rheumatol. 2023 Mar;42(3):879-888. doi: 10.1007/s10067-022-06389-4. Epub 2022 Oct 5. PMID 36197647